CLINICAL TRIAL: NCT05045118
Title: The Impact of Structured Patient Education Material (SPEM) in Improving Clinical and Behavioural Outcomes in Home-based Cardiac Rehabilitation Program Participants: A Pilot Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Malaya (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: MREC ID: 20201010-9146
Record Dates: First submitted 2021-09-01; First posted 2021-09-16 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: Ischaemic Heart Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention arm (Experimental): Single-arm prospective, multiple assessment intervention study. Participants will receive a digital structured patient education material
  Interventions: Other: Digital Structured Patient Education Material

INTERVENTIONS:
Other: Digital Structured Patient Education Material — Participants of home-based Cardiac Rehabilitation Program that are included in this research will be provided with a digital Structured Patient Education Material at the beginning of the program, and will be followed up for 12 weeks duration

SUMMARY:
This study aims to examine the impact of providing a digital education material to participants of home based cardiac rehabilitation in improving clinical and behavioural outcomes

DETAILED DESCRIPTION:
This is a pilot study aiming to assess the impact of providing a structured patient education material in a digital form to participants of home based cardiac rehabilitation program in University Malaya Medical Centre.

ELIGIBILITY:
Inclusion Criteria:

* Age 20-70 years
* Fulfills the low to moderate exercise participation risk criteria for Cardiac rehabilitation program phase 2 as per the American Association of Cardiovascular and Pulmonary Rehabilitation standards
* Able to participate in a treadmill exercise program
* Cognitively able to give consent, and able to read and utilize the digital education material

Exclusion Criteria:

* Stratified as high risk to participate in an aerobic exercise program as per the American Association of cardiovascular and Pulmonary Rehabilitation standards

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-03-30 (Actual); Primary Completion 2022-03-30 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Retention rate | 3 months
  The proportion of patients who completed the education material. The number of participants completed divided by the total number of participants, expressed in percentage
Cardiorespiratory fitness | 3 months
  Peak METs and HRmax measured by exercise stress testing, to estimate VO2 max. This measurement is recorded at pre and post 12 weeks of intervention

SECONDARY OUTCOMES:
Smoking status | 3 months
  Smoking status will be recorded as reported by patient upon recruitment, and at 1st, 2nd and 3rd month of program
Compliance to medication | 3 months
  Compliance to daily medication will be recorded as reported by patient upon recruitment, and at 1st, 2nd and 3rd month of program
Compliance to exercise | 3 months
  Number of hours of performing aerobic exercise per week upon recruitment, at 1st, 2nd, 3rd month

CONTACTS AND LOCATIONS:
Locations (1):
- University Malaya, Kuala Lumpur, Malaysia